CLINICAL TRIAL: NCT01778855
Title: An Ancillary Imaging Study to the Intravascular Cooling in the Treatment of Stroke 2 (ICTuS 2) Trial, an NIH-funded Project on the Safety and Efficacy of Hypothermia Combined With Thrombolysis
Brief Title: Hypothermia in Acute Stroke With Thrombolysis Imaging Evaluation of Revascularization
Acronym: HASTIER
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, David Liebeskind, Professor of Neurology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HASTIER; R01NS077706 (NIH)
Record Dates: First submitted 2013-01-23; First posted 2013-01-29 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Acute Ischemic Stroke
Keywords: stroke; hypothermia; thrombolysis; imaging; collateral circulation; recanalization; reperfusion
MeSH Terms: conditions — Ischemic Stroke; Stroke; Hypothermia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normothermia (Active Comparator): IV t-PA and normothermia
  Interventions: Other: IV t-PA and normothermia
- Hypothermia (Active Comparator): IV t-PA and hypothermia
  Interventions: Device: IV-tPA and hypothermia

INTERVENTIONS:
Other: IV t-PA and normothermia
  Other Names: t-PA as standard of care and normothermia
  Arms: Normothermia
Device: IV-tPA and hypothermia
  Other Names: Hypothermia is induced using the Celsius Control™ System and IV-tPA administered
  Arms: Hypothermia

SUMMARY:
The primary objective of this Phase 2 HASTIER study, as an ancillary study to ICTuS 2, is to compare key imaging measurements for serial changes in recanalization and reperfusion between hypothermia and normothermia treatment arms as intermediate outcomes of treatment effect. Secondary exploratory analyses include imaging of the neurovascular impact of reperfusion with hypothermia and tPA, including blood-brain barrier changes or permeability, hemorrhagic transformation, and infarct growth.

DETAILED DESCRIPTION:
A prospective imaging ancillary study coincides with recruitment of ICTuS 2 by using currently available imaging tools at a subset of multicenter sites. HASTIER will evaluate therapeutic response with imaging outcome measures for recanalization and reperfusion. Key scientific objectives include the evaluation of hypothermia on benchmark recanalization and reperfusion rates in 120 cases of middle cerebral artery (MCA) stroke. Recanalization will be measured with Thrombolysis in Myocardial Infarction (TIMI) score change from baseline-36 hour CT/MRI angiography. Reperfusion will be measured with Tmax > 6s lesion volume change from baseline-36 hour CT/MRI perfusion imaging. Secondary outcomes will be measured with serial changes in permeability abnormalities derived from CT/MRI perfusion imaging, hemorrhagic transformation, and infarct growth from baseline-36 hours. Correlation of these imaging parameters with clinical outcomes will provide insight to accelerate research during these translational steps in hypothermia treatment for acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for inclusion in the ICTuS 2/3 trial.
* Diagnosis of MCA stroke, confirmed by M1 or M2 proximal MCA occlusion on CT/MRI angiography.

Exclusion Criteria:

* Kidney dysfunction of such severity as to preclude routine administration of contrast media for CT/MRI angiography or perfusion imaging. Severe kidney dysfunction is defined by the American College of Radiology recommendations for use of contrast media.
* Known adverse reaction or allergy to such contrast media.

Ages: 22 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S Liebeskind, MD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Intercoastal Medical Group, Sarasota, Florida

REFERENCES:
- [Background] Lyden PD, Allgren RL, Ng K, Akins P, Meyer B, Al-Sanani F, Lutsep H, Dobak J, Matsubara BS, Zivin J. Intravascular Cooling in the Treatment of Stroke (ICTuS): early clinical experience. J Stroke Cerebrovasc Dis. 2005 May-Jun;14(3):107-14. doi: 10.1016/j.jstrokecerebrovasdis.2005.01.001. PMID 17904009
- [Background] Hemmen TM, Raman R, Guluma KZ, Meyer BC, Gomes JA, Cruz-Flores S, Wijman CA, Rapp KS, Grotta JC, Lyden PD; ICTuS-L Investigators. Intravenous thrombolysis plus hypothermia for acute treatment of ischemic stroke (ICTuS-L): final results. Stroke. 2010 Oct;41(10):2265-70. doi: 10.1161/STROKEAHA.110.592295. Epub 2010 Aug 19. PMID 20724711

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normothermia | Hypothermia
Started | 2 | 4
Completed | 2 | 3
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normothermia | Hypothermia | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recanalization
Description: To determine whether hypothermia alters recanalization with standard thrombolytic treatment with intravenous (IV) tissue plasminogen activator (tPA) for acute ischemic stroke in humans. The hypothesis is that hypothermia does not impair recanalization (opening of the artery). Recanalization will be measured with Thrombolysis in Myocardial Infarction (TIMI) score change from baseline angiography to 36 hour angiography. TIMI is cored per published definition.
  Additional data for secondary analyses were not acquired to permit analyses.
Time Frame: 36 hours
Population: Recanalization at 36 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Normothermia | Hypothermia
Number analyzed (Participants) | 2 | 4
Participants | 2 | 3

ADVERSE EVENTS:
Arm/Group | Normothermia | Hypothermia
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normothermia (N=2) | Hypothermia (N=4)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Death (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Normothermia (N=2) | Hypothermia (N=4)
Abnormal coagulation profile (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aspiration pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral edema (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Elevated troponin (Cardiac disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Fluid overload (Vascular disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pain (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Topical fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of ancillary study leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No